CLINICAL TRIAL: NCT04865432
Title: Evaluating the Effect of Solius UV Light Source in Improving Serum Levels of 25-hydroxyvitamin D in Vitamin D Deficient/ Insufficient Adults of Various Skin Types: A Feasibility Study
Brief Title: Solius UV Light Source in Improving Serum Levels of 25-hydroxyvitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-41681
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Vitamin D Deficiency; Vitamin D Insufficiency
Keywords: Vitamin D; Ultraviolet B radiation
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- UVB treatment (Experimental): Participants will first undergo an evaluation of each individual's sensitivity to the Solius Photobiological System UVB using the device titration system for the first 5 weeks. Once determined, participants will participate in a 4-week intervention where they will be exposed to their individualized titration evaluation.
  Interventions: Device: UVB treatment

INTERVENTIONS:
Device: UVB treatment — 5 weeks of UVB titration to determine individual's UVB sensitivity followed by 4 weeks of UVB exposure intervention

SUMMARY:
This is a feasibility interventional study seeking to determine the safety and efficacy of the Solius Photobiologic System in increasing the serum levels of 25(OH)D in a vitamin D deficient/insufficient adult population.

DETAILED DESCRIPTION:
The investigators will conduct an interventional study to determine the changes in the changes in serum 25-hydroxyvitamin D levels between subjects who receive weekly exposures to Ultraviolet B Radiation (UVB) generated by the Solius Photobiological System for 4 weeks. Subjects will first undergo an evaluation of each individual's sensitivity to the Solius Photobiological System UVB using the device titration system for the first 5 weeks. Once determined after the 5 weeks, the subjects will be enrolled in a 4-week study where they will be exposed to their individualized titration evaluation. Approximately 14 adult participants will be enrolled for serum 25-hydroxyvitamin D screening. The investigators expect to enroll 10 vitamin D-deficient or insufficient subjects in this study. Serum 25-hydroxyvitamin D levels will be measured prior to the first titration (week 2), prior to the intervention (week 6) and after the end of the study, and and the changes in serum 25-hydroxyvitamin D levels will be analyzed. The investigators expect that the levels will increase from the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 22 years old
2. Male or Female
3. Skin Type I-VI
4. Women of childbearing potential must be on birth control and not pregnant based on a negative pregnancy test at baseline.
5. Ability and Willingness to give informed consent and comply to protocol requirements
6. Serum total 25(OH)D < 30 ng/mL

Exclusion Criteria:

1. Ongoing treatment with supplemental or pharmacological doses of vitamin D, vitamin D metabolites or analogues
2. Pregnant
3. History of underlying photosensitivity
4. Use of medications that cause a photosensitivity reaction (including but not limited to): tetracycline, tretinoin, amiodarone, doxycycline, naproxen, diphenhydramine, methotrexate, and hydrochlorothiazide
5. History of skin cancer
6. Plan to received significant sun exposure below the 33rd parallel during study
7. Used tanning or phototherapy devices within the last 30 days
8. Vitamin D supplement use of more than 600 IUs daily.
9. Systemic steroids use
10. H1 antihistamine use in the last 7 days
11. Diagnosed with light allergies (including but not limited to): actinic prurigo, polymorphous light eruption, or solar urticaria
12. Diagnosed with light sensitivities (including but not limited to): protoporphyria, photodermatitis, xeroderma pigmentosum, lupus erythematosus, chronic actinic dermatitis, or UV-sensitive syndrome

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holick, PhD MD, Principal Investigator — Boston University
Locations (1):
- General Clinical Research Unit (GCRU) BU School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- UVB Treatment: Participants will first undergo an evaluation of each individual's sensitivity to the Solius Photobiological System Ultraviolet B (UVB) using the device titration system for the first 5 weeks. Once determined, participants will participate in a 4-week intervention where they will be exposed to their individualized titration evaluation.
Period: Overall Study
Arm/Group | UVB Treatment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | UVB Treatment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Serum 25-hydroxyvitamin D level [Mean (Standard Deviation); unit: ng/ml] | 24.0 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Serum 25-hydroxyvitamin D
Description: Serum 25-hydroxyvitamin D level at 4 weeks of intervention (the end of study)
Time Frame: Serum 25-hydroxyvitamin D at 4 weeks of intervention
Measure: Mean (Standard Deviation); unit: ng/nl
Arm/Group | UVB Treatment
Number analyzed (Participants) | 10
ng/nl | 25.4 (7.3)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | UVB Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04865432/Prot_SAP_000.pdf